CLINICAL TRIAL: NCT00662883
Title: A Randomized, Open Label Study to Assess the Effects of a Nasal Corticosteroid on the Pharmacokinetics, Safety, and Tolerability of PMI-150 (Intranasal Ketamine Hydrochloride) 30 mg
Brief Title: Assessing the Effects of a Nasal Corticosteroid on PMI-150 (Intranasal Ketamine)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Javelin Pharmaceuticals, Inc., Javelin Pharmaceuticals, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: KET-PK-009
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Healthy
Keywords: ketamine; corticosteroid; intranasal; phase I; Healthy volunteers
MeSH Terms: interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): * PMI-150 (intranasal ketamine HCl), day 1
  * mometasone furoate, days 2-15
  * PMI-150 (intranasal ketamine HCl), day 15
  Interventions: Drug: PMI-150 (intranasal ketamine HCl); mometasone furoate

INTERVENTIONS:
Drug: PMI-150 (intranasal ketamine HCl); mometasone furoate — * 1 dose PMI-150 (intranasal ketamine HCl); day 1
  * mometasone furoate, daily; days 2-15
  * 1 dose PMI-150 (intranasal ketamine HCl); day 15
  Other Names: Nasonex

SUMMARY:
To assess the effects of nasal corticosteroid treatment on the rate and extent of intranasal absorption of PMI-150 (intranasal ketamine HCl)

DETAILED DESCRIPTION:
Subjects will participate in a two-period, single-sequence study to assess the effects of administration of a nasal corticosteroid, Nasonex (mometasone furoate), on the pharmacokinetics, safety and tolerability of PMI-150 (intranasal ketamine HCl) in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* nonsmoker
* no drug use

Exclusion Criteria:

* nasal abnormalities
* airway abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Javelin Pharmaceuticals, Inc, Study Director — Javelin Pharmaceuticals
Locations (1):
- Baltimore, Maryland, United States